CLINICAL TRIAL: NCT02631629
Title: Food-based Solutions for Optimal Vitamin D Nutrition and Health
Acronym: ODIN_FOOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Denmark (Other)
Collaborators: Seventh Framework Programme (Other)
Responsible Party: Principal Investigator, Inge Tetens, Professor, Technical University of Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-15008276; FP7-613977-ODIN (Other Grant/Funding Number: EU FP7)
Record Dates: First submitted 2015-11-11; First posted 2015-12-16 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D; Fortification
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Food, Fortified

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Non-fortified foods SA (Placebo Comparator): Non-fortified foods (eggs, cheese, yoghurt, crips bread) (placebo), women of South Asian (SA) origin
  Interventions: Other: Non-fortified foods
- Non-fortified foods CA (Placebo Comparator): Non-fortified foods (eggs, cheese, yoghurt, crips bread) (placebo), women of Caucasian (CA) origin
  Interventions: Other: Non-fortified foods
- Vitamin D fortified foods SA (Active Comparator): Vitamin D fortified foods (eggs, cheese, yoghurt, crips bread), women of South Asian (SA) origin
  Interventions: Other: Fortified foods
- Vitamin D fortified foods CA (Active Comparator): Vitamin D fortified foods (eggs, cheese, yoghurt, crips bread), women of Caucasian (CA) origin
  Interventions: Other: Fortified foods

INTERVENTIONS:
Other: Non-fortified foods — The non-fortified placebo foods are eggs, cheese, yoghurt and crisp bread (without vitamin D added).
  Arms: Non-fortified foods CA; Non-fortified foods SA
Other: Fortified foods — The fortified intervention foods are eggs, cheese, yoghurt and crisp bread (with about 20 mcg/day).
  Arms: Vitamin D fortified foods CA; Vitamin D fortified foods SA

SUMMARY:
This project aims at proving the efficacy and safety of food based solutions to prevent vitamin D deficiency in high risk populations of Caucasian and South Asian origin living in Denmark.

DETAILED DESCRIPTION:
The study is a 12 week double-blinded, randomised, placebo-controlled food-based intervention trial in a real-life setting. 140 (18-50 y) women in risk of vitamin D deficiency and with Caucasian or South Asian origin. The two ethnic groups of women will each be randomised into two groups. One receiving vitamin D fortified foods and the other receiving the same kind of foods non-fortified. Foods given in the study period are free of charge for the participants and will be handed out every second week. The foods are eggs, yoghurt, cheese and crisp bread.

The study includes a baseline visit and a final visit, at both visits blood samples will be drawn, anthropometrics, muscle strengths, dietary and background questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 year old women
* Low consumption of fish and fish products
* Low intake of vitamin D containing supplements
* No use of sunning facilities
* No planned sun-holiday between October 2015 and May 2016

Exclusion Criteria:

* Pregnancy and breastfeeding
* Menopause
* Serious diseases (cancer, server liver or kidney insufficiencies, sarcoidosis and other granulomatous diseases) and medicines affecting the vitamin D metabolism (steroids, antiepileptic, thyroid hormones, bisphosphonates, oestrogen).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 143 (Actual)
Dates: Start 2015-11; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
The change in vitamin D status measured as serum 25-hydroxyvitamin D | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Inge Tetens, Professor, Principal Investigator — Technical University of Denmark
Locations (1):
- Technical University of Denmark, Søborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gronborg IM, Tetens I, Christensen T, Andersen EW, Jakobsen J, Kiely M, Cashman KD, Andersen R. Vitamin D-fortified foods improve wintertime vitamin D status in women of Danish and Pakistani origin living in Denmark: a randomized controlled trial. Eur J Nutr. 2020 Mar;59(2):741-753. doi: 10.1007/s00394-019-01941-6. Epub 2019 Mar 9. PMID 30852657